CLINICAL TRIAL: NCT04815070
Title: Comparison of Fasting Gastric Volume Using Ultrasound in Diabetic and Non-Diabetic Elderly Patients Undergoing Staged Bilateral Total Knee Arthroplasty: A Prospective Observational Study
Brief Title: Gastric Volume in Diabetic Patients Undergoing Staged Bilateral Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2103/673-307
Record Dates: First submitted 2021-03-22; First posted 2021-03-24 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Degenerative Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diabetic: A group of diabetic patients who have fasted for at least 8 hours undergoing staged bilateral total knee arthroplasty.
  Interventions: Procedure: Ultrasonic measurement of antral area
- Non-Diabetic: A group of non-diabetic patients who have fasted for at least 8 hours undergoing staged bilateral total knee arthroplasty.
  Interventions: Procedure: Ultrasonic measurement of antral area

INTERVENTIONS:
Procedure: Ultrasonic measurement of antral area — Ultrasound exam is done before the induction of spinal anesthesia. Three consecutive measurements of the anteroposterior (AP) and cranio-caudal (CC) diameters are performed.
  The cross-sectional area (CSA) of antrum is shown by the following formula: CSA = AP x CC x ㅠ/4.
  Antral area will correspond to the average of the three measures.

SUMMARY:
Aspiration of gastric contents during perioperative period is a grave complication with significant morbidity and mortality. Diabetic patients have a higher incidence of autonomic dysfunction, causing gastropathy. They are known to have gastroparesis and the consequent delayed gastric emptying which predisposes them to an increased risk of aspiration than the general population. Furthermore, other common factors can influence the gastric emptying rate, as for example, old age, pain, and the use of opioid analgesics.

In the previous study, evidence of increased pain was reported in patients undergoing staged bilateral total knee arthroplasty, in whom the second operated knee had greater sensitivity (tertiary hyperalgesia) due to the surgical injury to the first operated knee.

In the present study, we will evaluate the effect of old age, diabetes, surgical stress, pain, and the use of analgesics on the residual gastric volume in elderly patients undergoing staged-bilateral total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for staged bilateral total knee arthroplasty aged 65 to 85 years
* American Society of Anestheiologist physical status classification 1, 2, and 3
* Body mass index < 35 kg/cm2

Exclusion Criteria:

* Previous surgery of the upper gastrointestinal tract
* Achalasia

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Study participants will be patients whom are scheduled to undergo staged bilateral total knee arthroplasty requiring preoperative fasting period of at least 8 hours. 40 patients will be recruited in total. One cohort consisting 20 patients will be diabetic. The other cohort consisting of 20 patients will be non-diabetic.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Volume of Gastric Contents | Less than one hour prior to surgery
  A "full stomach" is defined as on containing a) solid or thick fluid content or b) 1.5 mL/kg of clear fluid.

SECONDARY OUTCOMES:
Numerical rating pain scale | One hour prior to surgery, Postoperative 24 and 48 hour
  Postoperative pain score (0 = no pain, 10 = very severe pain)
Rescue analgesics | Postoperative 24 and 48 hour
  Amounts of the analgesics administered to manage the postoperative pain

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No